CLINICAL TRIAL: NCT04089969
Title: Cardiac Risk Assessment Using Standard of Care Versus CTA and Heart Flow FFRct in Patients With End-Stage Liver Disease Under Consideration for Liver Transplant.
Brief Title: Cardiac Risk Assessment Using Standard of Care Versus CTA and Heart Flow FFRct
Acronym: CRASCH-Liver
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Essential staff for study execution left the institution and no suitable replacement could be found.
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Robert Safian, MD., Corewell Health East
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-151
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Acute Liver Failure; Liver Transplant
Keywords: CTA, FFRct, CAD; End Stage Liver DIsease; Liver failure, Liver transplant
MeSH Terms: conditions — Coronary Artery Disease; Liver Failure, Acute; End Stage Liver Disease; Liver Failure

STUDY DESIGN:
Intervention Model Description: Single-Blind decision-making study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Evaluation of Standard of care followed by CTA/FFRct (Experimental): Patient received clinical recommendation based on the Standard of Care i.e 2 D echocardiogram, plus ECG, plus, pharmacological stress test followed by re-evaluation of clinical recommendation with addition of CTA/FFRct
  Interventions: Diagnostic Test: CTA/FFRct; Diagnostic Test: SOC cardiovascular evaluation

INTERVENTIONS:
Diagnostic Test: CTA/FFRct — Computed Tomography Angiogram with Fractional Flow Reserve. A Ct scan of the heart's blood vessels.
Diagnostic Test: SOC cardiovascular evaluation — Standard of care (SOC) cardiovascular evaluation i.e ECG, 2 D echocardiogram and pharmacologic stress test such as Dobutamine and Myocardial Perfusion Imaging stress test.

SUMMARY:
Coronary Artery Disease (CAD) is the narrowing or blockage of the artery of the heart and is prevalent in end-stage liver disease. Consultation with cardiologist and stress tests are recommended to patients under consideration for liver transplant. The purpose of this study is to evaluate if Computed Tomography Angiogram (CTA) and CTA-derived Fractional Flow Reserve (FFRct) procedure influences decisions about further cardiac testing compared with Standard of Care (SOC) such as consultation by a cardiologist, Echocardiogram (ultrasound of the heart), Electrocardiogram (ECG) and stress tests.

DETAILED DESCRIPTION:
The purpose of this study is to determine in end-stage liver disease patients whether non-invasive assessment of coronary artery disease prior to liver transplant using CTA (CTA) and CTA-derived Fractional Flow Reserved (FFRct) is superior to current standard of care (SOC) cardiovascular evaluation such as formal consultation by a cardiologist, electrocardiogram, echocardiogram, and pharmacological stress test such (e.g. Dobutamine stress echocardiogram and lexiscan myocardial perfusion imaging). The investigational portion of this study is the CTA and FFRct, which is a special x-ray scan that can identify blockages in the arteries and determine if blood flow is impaired. The CTA and FFRct will be done within 2 weeks after the standard of care evaluation.

All 100 patients will undergo standard of care stress test plus CTA/FFRct. The referring cardiologist will be blinded to the results of CTA/FFRct, and will make an "initial" recommendation based on the standard of care evaluation. After making the "initial" recommendation, the referring cardiologist will be unblinded to the CTA/FFRct results and make a "final" recommendation. The "initial" recommendation will consist of one of the following: further cardiac evaluation is not needed or cardiac catheterization is required. The "final" recommendation will consist of one of the following: further cardiac evaluation is not needed or cardiac catheterization is required. All patients will receive a 1 year phone follow up call.

The hypothesis is that in End Stage Liver Disease (ESLD) patients, non-invasive assessment for CAD using CTA/FFRct is superior to SOC cardiovascular evaluation (stress etst, echocardiogram, ECG). This study will look at the frequency of how often CTA/FFRct changed the clinical recommendation compared with the standard of care alone (Initial recommendation versus final recommendation).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end-stage liver disease
2. Patients undergoing cardiovascular risk assessment prior to liver transplantation -

Exclusion Criteria:

1. Estimated Glomerular Filtration Rate (eGFR) < 30 cc/min/1.73 m^2 (unless patient is on dialysis or renal transplant is planned)
2. Heart rate > 90 bpm despite beta blocker therapy
3. Body Mass Index (BMI) > 40 plus chest obesity (i.e. truncal obesity and normal chest morphology is not an exclusion)
4. Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in clinical recommendation | within 2 weeks after SOC assessment
  Number of Participants whose clinical recommendation as initially determined by SOC assessment is changed following CTA/FFRct assessment.

SECONDARY OUTCOMES:
Frequency of detecting Coronary Artery Disease (CAD) by CTA/FFRct | within 2 weeks after SOC assessment
  Number of Participants with agreement in CAD status detected by both Pharmacological stress test and also CTA/FFRct.
Cardiovascular morbidity | 1 year
  Number of participants with cardiovascular related Death, Myocardial Infarction (MI: defined as any 2 of following; 1. ischemic chest pain, 2. elevated troponin 3. pathologic Q waves or ischemic ST changes), or ischemia driven revascularization
Projected Health Care Cost | within 2 weeks after SOC assessment
  Dollar value of Standard of care treatment (related to CAD) and CTA/FFRct
Frequency of Detecting Myocardial Ischemia and the frequency of detecting the correct territory of the Myocardial Ischemia. | within 2 weeks after SOC assessment
  Number of participants with Myocardial Ischemia and correct territory of Myocardial Ischemia detected by Pharmacological Stress Test vs CTA/FFRct

CONTACTS AND LOCATIONS:
Overall Officials: Robert Safian, MD, Principal Investigator — Corewell Health East

IPD SHARING:
Plan to Share IPD: No